CLINICAL TRIAL: NCT03177369
Title: Teicoplanin-based Antimicrobial Therapy in Staphylococcus Aureus Bone and Joint Infection: Tolerance, Efficacy and Experience With Subcutaneous Administration
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0385
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Teicoplanin-based Antimicrobial Therapy; Staphylococcus Aureus; Bone and Joint Infection
Keywords: Bone and joint infection; Staphylococcus aureus; Teicoplanin; Subcutaneous administration
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Staphylococci represent the first etiologic agents of bone and joint infection (BJI), leading glycopeptides use, especially in case of methicillin-resistance or betalactam intolerance. Teicoplanin may represent an alternative to vancomycin because of its acceptable bone penetration and possible subcutaneous administration. Various studies have shown that teicoplanin pharmacodynamic profile was superior compared to vancomycin regarding bone diffusion. Few studies have investigated the use of teicoplanin in BJI, particularly through subcutaneous administration.

The aim of this study assesses the efficacy and tolerance of teicoplanin in S. aureus BJI, especially focusing on subcutaneous use. This study is a retrospective single-center observational cohort study (2001 to 2011) including all consecutive patients managed at our institution receiving teicoplanin as part of S. aureus BJI treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients with bone and joint infection caused by S. aureus receiving teicoplanin (IV or SC) as part to treat the infection

Exclusion Criteria:

- Patients with diabetic foot- and decubitus ulcer-related BJI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bone and joint infection caused by S. aureus managed in the reference center for BJI in Lyon, between 2001 and 2011.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of teicoplanin in S.aureus bone and joint infection | 90 weeks
  The median total duration of follow-up is 90 weeks. Outcome of patients having had teicoplanin is described in this part. Treatment failure is defined as persisting infection under appropriate antimicrobial therapy, relapse after the interruption of antimicrobial therapy, necessity of surgical revision on the account of persisting septic focus ≥5 days after the first intervention, superinfections, and/or fatal outcome if BJI-related.
  The results obtained with IV or SC administration are compared.

SECONDARY OUTCOMES:
Tolerance of teicoplanin in S.aureus bone and joint infection | 6 weeks
  The median total duration of teicoplanin therapy is 6 weeks (IV or SC). Teicoplanin-related adverse events (AE) occurring during follow-up are notified and classified according to the Common Terminology Criteria for Adverse Events (CTCAE, National Cancer Institute, 2003). Teicoplanin accountability in the AE occurrence is left to the clinician appreciation, with the help of a pharmacovigilance specialist in doubtful cases.
  The results obtained with IV or SC administration are compared.
Pharmacocinetiks characteristics : Cmin value | 2 weeks
  During the first 14 days of treatment, at least one Cmin value is available. A Cmin >15 mg/L is taken as an acceptable therapeutic target. Patients with a Cmin >25 mg/L is considered as overexposure.
  (The results for overexposure and Cmin under the therapeutic target are compared for IV and SC administration.)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse - Centre de reference des infection ostéo-articulaires de Lyon, Lyon, France